CLINICAL TRIAL: NCT06531291
Title: Surufatinib Combined With Serplulimab and Standard Chemotherapy as First-line Treatment in Advanced Solid Tumors With Neuroendocrine Differentiation: A Single-arm, Multi-cohort, Open-label, Single-center, Prospective, Exploratory Clinical Study
Brief Title: Surufatinib Combined With Serplulimab and Standard Chemotherapy as First-line Treatment in Advanced Solid Tumors With Neuroendocrine Differentiation
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, liwei wang, Director of department of oncology, RenJi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPOGCNED-14
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: ESCC; Biliary Tract Cancer; Gastric Cancer; Pancreas Cancer
Keywords: surufatinib; Neuroendocrine Differentiation
MeSH Terms: conditions — Biliary Tract Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms | interventions — surufatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surufatinib + serplulimab + standard chemotherapy (Experimental)
  Interventions: Drug: Surufatinib; Drug: Serplulimab; Drug: standard chemotherapy

INTERVENTIONS:
Drug: Surufatinib — 250 mg, po, qd, q3w
Drug: Serplulimab — 200 mg, iv, d1, q3w
Drug: standard chemotherapy — Decided by PI

SUMMARY:
Currently, there are no standard treatment and relevant exploration for solid tumors patients with NED. The study aims to explore the efficacy and safety of surufatinib combined with serplulimab and standard chemotherapy in the treatment ofadvanced solid tumors with NED, in order to provide a new treatment option for advanced solid tumors patients with NED.

DETAILED DESCRIPTION:
This is a single-arm, multi-cohort, open-label, single-center, prospective, exploratory clinical study. We planned to enroll 80 patients who would receive surufatinib plus tislelizumab until disease progression, intolerance, or withdrawal of consent. The study aims to explore the efficacy and safety of surufatinib combined with serplulimab and standard chemotherapy in the treatment of advanced solid tumors with NED, in order to provide a new treatment option for advanced solid tumors patients with NED.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed locally advanced or metastatic unresectable ESCC, BTC, PC or GC with an abnormal NED or NE phenotype (without neuroendocrine morphologic features and positive immunohistochemical expression of at least one neuroendocrine marker (CgA, Syn));
* Have at least one measurable lesion according to RECIST v1.1;
* ECOG performance status: 0-1;
* No previous systemic therapy;
* Urine protein< ++ . If Urine protein ≥ ++ ,the amount of urine protein in 24 hours ≤1.0g;
* Expected survival time > 3 months;

Exclusion Criteria:

* Have uncontrolled hypertension, defined as systolic blood pressure >150 mmHg or diastolic blood pressure >90 mm Hg, while under anti-hypertension treatment;
* With active bleeding or bleeding tendency;
* Severe history of cardiovascular and cerebrovascular diseases;
* Other malignancies diagnosed within the previous 5 years, except basal cell carcinoma or cervical carcinoma in situ after radical resection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2027-08-09 (Estimated); Study Completion 2027-08-09 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | approximately 1 years
  time from first-dose to the first documented disease progression or death

SECONDARY OUTCOMES:
Objective response rate (ORR) | approximately 1 years
  the proportion of patients with complete response or partial response, using RESIST v1.1
Disease Control Rate (DCR) | approximately 1 years
  the proportion of patients with complete response, partial response or stable disease, using RESIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Liwei Wang, Doctorate, Principal Investigator — RenJi Hospital
Locations (1):
- Renji hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No